CLINICAL TRIAL: NCT02760160
Title: Dietary Prevention of Photodamage in Skin With Grapes: A Human Clinical Study
Brief Title: Dietary Prevention of Photodamage in Skin With Grapes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Craig Elmets, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F140627004
Record Dates: First submitted 2015-12-17; First posted 2016-05-03 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2018-01

CONDITIONS: Non-melanoma Skin Cancer
MeSH Terms: interventions — whole grape extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reconstituted grape powder (Other): Open grape powder pouch and pour contents into volumetric measuring device. Add approximately 180 mL of water to container with grape powder. Stir for a minimum of 30 seconds and ingest.
  Interventions: Other: Reconstituted grape powder

INTERVENTIONS:
Other: Reconstituted grape powder — To prevent UV-induced skin cancers. Each subject's will have one arm exposed to 6 separate doses of UV (J/m2) [114, 217, 343, 500, 619, 848].
  Other Names: Grape powder

SUMMARY:
To assess the effect of orally administered grape powder on the sunburn reaction in humans.

DETAILED DESCRIPTION:
To determine whether oral grape powder will result in a reduction in biomarkers associated with basal cell carcinomas (BCCs) and squamous cell carcinomas (SCCs). Biomarkers taken from non-sun-exposed skin and UV-exposed skin before and after treatment will be compared.

The ultimate goal of this study will be to generate new knowledge of the photoprotective effect of grape powder on UV exposure. The results may be employed as the basis for a larger clinical trial to evaluate the potential of grapes to prevent non-melanoma skin cancers (NMSCs) and sun damage.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 and older
* Patient able to understand requirements of the study and risks involved
* Patient able to sign a consent form

Exclusion Criteria:

* Patients Fitzpatrick IV-VI
* A recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation
* A known history of photosensitivity disorders
* A known history of melanoma or non-melanoma skin cancers
* Those planning on going to the tanning parlors
* Using any of the photosensitizing medication
* A woman who is lactating, pregnant, or planning to become pregnant
* Patient planning on exposing the irradiated or control areas to the sun

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting protective effect against sunburn response to UVG and/or UVA1 following administration of dietary grape powder. | 2 weeks
  Assessment will be quantified by evaluation of a person's minimal erythema dose (MED), the smallest amount of ultraviolet (UV) required to achieve a sunburn response. 6 small areas of skin (2 inches by 2 inches) on the inner part of a person's arm will be exposed to 6 separate but increasing doses of UV. 24 hours after UV treatment, the area that received the smallest dose of UV and has a visible area of redness will be marked and the respective UV dose will be considered the MED. A desirable outcome would be if an individual's MED goes up after 2 weeks of grape treatment.

SECONDARY OUTCOMES:
Measure whether dietary grape powder results in a significant (p<0.05 using parire ttest) % change in markers associated with NMSC as measured by it biomarker: ornithine decarboxylase (ODC) | 2 weeks
  Immunohistochemistry (IHC) will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated.
Measure whether dietary grape powder results in a significant (p<0.05 using parire ttest) % change in markers associated with NMSC as measured by it biomarker: proliferating cell nuclear antigen (PCNA) | 2 weeks
  Immunohistochemistry (IHC) will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: Ki67 | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: Cyclin D1 | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: Cyclooxygenase-2 (COX-2) | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: matrix metalloproteinase-7 (MMP-7) | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated.
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: matrix metalloproteinase-9 (MMP-9) | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: Normal p53 | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated.
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: Mutant p53 | 2 weeks
  IHC will be used to quantify the percentage of stained cells using the microscope. This percentage will be compared in biopsy samples before and after grape treatment for each individual. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of stained cells)/(total number of patients). Furthermore, western blot will be used to quantify the level of protein expression. The expression of each marker will be compared in each patient and the aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in expression of the respective biomarker)/(total number of patients). The percent change of each biomarker expression before and after treatment if a notable difference is observed using either IHC or western blot, or both will be calculated.
Determine whether dietary grape powder has photoprotective activities over a period of 2 weeks and resulting in a significant change in biomarkers associated with NMSC as measured by biomarker: Sunburnt cells | 2 weeks
  Routine histology (hematoxylin and eosin stain) will be used and the number of sunburnt cells will be quantified under the microscope. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of sunburnt cells)/(total number of patients). We will also calculate the change in the number of sunburnt cells before and after treatment if a notable difference is observed.
Determine whether dietary grape powder has photoprotective activities resulting in a significant change in biomarkers associated with NMSC: by biomarker: Terminal deoxynucleotidyl transferase dUTP nick end labeling (TUNEL)-positive cells | 2 weeks
  The number of TUNEL-positive cells, which will be fluorescent, will be quantified under the microscope. The aggregate data will be presented using the following formula: (number of patients with a statistically significant decrease in the percentage of TUNEL-positive cells)/(total number of patients). We will also calculate the percent change TUNEL-positive cells before and after treatment if a notable difference is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Elmets, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Dermatology, Birmingham, Alabama, United States